CLINICAL TRIAL: NCT03377374
Title: Randomized Controlled Trial on the Safety and Efficacy of L. Reuteri ATCC PTA 5289 & L. Reuteri DSM 17938 for the Treatment of Children With Pharyngitis and/or Tonsillitis: A Proof of Concept
Brief Title: L. Reuteri ATCC PTA 5289 & L. Reuteri DSM 17938 for the Treatment of Children With Pharyngitis and/or Tonsillitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, Head of Research on Translational Research Center on Mother-Child Health, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB0140
Record Dates: First submitted 2017-11-29; First posted 2017-12-19 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Pharyngitis; Tonsillitis
MeSH Terms: conditions — Pharyngitis; Tonsillitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, double blind allocation concealment, parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization list will by assembled by independient organization not related with participant, care provider, investigators or sponsors. eCRF will include randomization selection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): L. reuteri ATCC PTA 5289 + L. reuteri DSM 17938 at a dose of 2x10^8 Colony Forming Units (CFU)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Five drops of Placebo taken twice a day (in the morning and in the evening).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — L. reuteri Prodentis oil drops (L. reuteri DSM 17938 and L. reuteri ATCC PTA 5289) will be given at a dose of 2x108 Colony Forming Units (CFU). Five drops are to be taken twice a day (in the morning and in the evening) giving a daily dose of 4x108 CFU/day.
  Arms: Probiotic
Other: Placebo — Five drops of Placebo taken twice a day (in the morning and in the evening).
  Arms: Placebo

SUMMARY:
RCT in children (6m to 5y) with pharyngitis and/or tonsillitis who will be allocated to receive for 10 days L. reuteri DSM 17938 + L. reuteri ATCC PTA 5289) at a dose of 2x10^8 Colony Forming Units (CFU). Five drops are to be taken twice a day (in the morning and in the evening) or placebo drops, as treatment for clinical condition. Duration of symptoms and reduction of pain (odynophagia) severity during treatment will be measured as primary outcome

DETAILED DESCRIPTION:
Rationale. Acute respiratory infections (ARIs) are a common problem in the first decade of life. The yearly prevalence of respiratory tract infections in an otherwise healthy 3-year old child is about three to 10 infections. Children between 6 months and 5 years are more prone to develop pharyngitis and tonsillitis compared to older children. 60-70% of children with F/T lies within this age group. Aetiology the pharyngitis and tonsillitis is viral in 70% of all cases In developing countries 6/10 cases are treated using antibiotics, regardless of clinical guidelines or standard of care documents recommending only to use symptomatic drugs (NSAID).

Primary outcome. Duration of symptoms and reduction of pain (odynophagia) severity Secondary outcomes. Days with fever secondary to RTIs; Number of children receiving antibiotic treatment in each treatment group; Days of medical office visits or emergency visits; Total amount of medical office visits or emergency visits during the study, secondary to episodes of RTI; Days of absences from day care centre; Direct and Indirect costs Total costs of treatments including visit to private office, visit to emergency department, cost of treatment (NSAIDs + Probiotics vs NSAIDs + Placebo); Frequency of adverse events; Viral/bacterial load (multiplex-PCR); IgA in saliva and Change in salivary inflammatory biomarkers.

Interventions. L. reuteri DSM 17938 + L. reuteri ATCC PTA 5289) will be given at a dose of 2x10^8 Colony Forming Units (CFU). Five drops are to be taken twice a day (in the morning and in the evening) giving a daily dose of 4x108 CFU/day. The placebo drops will have identical ingredients except for lacking the bacteria. Five drops are to be taken twice a day (in the morning and in the evening).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Infants suffering from pharyngitis and/or tonsillitis
* Born at term (36 weeks of gestation)
* Any gender
* 6 months to 5 years old
* Birth weight >2500 g
* Same socioeconomic background
* Written informed consent from at least one parent or legal guardian

Exclusion Criteria:

* Use of antibiotics or probiotic products 2 weeks' prior inclusion in the study
* Eight or more new ear infections (otitis media) within 12 months
* Two or more serious sinus infections within 12 months
* Two or more episodes of pneumonia within 12 months
* Two or more invasive infections in the history (meningitis, cellulitis, osteomyelitis, septicaemia)
* Failure to gain weight or grow normally
* Chronic diarrhoea
* Recurrent deep skin or organ abscesses,
* Persistent superficial candidiasis after 1 year of age
* Use of two or more months on antibiotics for respiratory infections on the last year before considered eligible
* Gastroesophageal reflux
* Allergy
* Asthma
* A1-antitrypsin deficeincy
* Primary or secondary ciliary dyskenisia
* Congenital anomalies of respiratory tract
* Supplementation of probiotics 2 weeks before inclusion in the study and during the whole study period
* If the mother is breastfeeding the child participating in the trial the mother should not use supplementation of probiotics 2 weeks before and during the study period
* Concurrent participation in other clinical trials

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement | 10 days
  Duration of respiratory symptoms

SECONDARY OUTCOMES:
Fever improvement | 10 days
  Total number of hours during the study that the child is with temperature >37.5oC measured twice a day since the moment they start to use the interventions and until the last visit into the study
Use of antibiotics | 10 days
  Total amount of days of antibiotic use during the study, secondary to the presence of episodes of RTI, reported since the beginning of the study products administration until the last visit occur
Medical/Emergency visits | 10 days
  Total amount of medical office visits or emergency visits during the study, secondary to episodes of RTI, reported since the beginning of the study products administration until the last visit occurs
Abseentisim | 10 days
  Total amount of days of absences from the day care centre during the study, secondary to the presence of episodes of RTI, reported since the beginning of the study products administration until the last visit occurs.
Costs of intervention | 10 days
  Total costs of treatments including visit to private office, visit to emergency department, cost of treatment (NSAIDs + Probiotics vs NSAIDs + Placebo)
Adverse events | 10 days
  Total number of adverse events which be reported by parents starting after randomization and finishing at the moment of last visit
Inflammatory improvements | 10 days
  Changes in IgA in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gutierrez Castrellon, MD, MSc, DSc, Principal Investigator — Innovacion y Desarrollo de Estrategias en Salud
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laursen RP, Larnkjaer A, Ritz C, Hauger H, Michaelsen KF, Molgaard C. Probiotics and Child Care Absence Due to Infections: A Randomized Controlled Trial. Pediatrics. 2017 Aug;140(2):e20170735. doi: 10.1542/peds.2017-0735. Epub 2017 Jul 3. PMID 28674113
- [Result] Gerasimov SV, Ivantsiv VA, Bobryk LM, Tsitsura OO, Dedyshin LP, Guta NV, Yandyo BV. Role of short-term use of L. acidophilus DDS-1 and B. lactis UABLA-12 in acute respiratory infections in children: a randomized controlled trial. Eur J Clin Nutr. 2016 Apr;70(4):463-9. doi: 10.1038/ejcn.2015.171. Epub 2015 Oct 14. PMID 26463725
- [Result] Taipale TJ, Pienihakkinen K, Isolauri E, Jokela JT, Soderling EM. Bifidobacterium animalis subsp. lactis BB-12 in reducing the risk of infections in early childhood. Pediatr Res. 2016 Jan;79(1-1):65-9. doi: 10.1038/pr.2015.174. Epub 2015 Sep 15. PMID 26372517
- [Result] Maldonado J, Canabate F, Sempere L, Vela F, Sanchez AR, Narbona E, Lopez-Huertas E, Geerlings A, Valero AD, Olivares M, Lara-Villoslada F. Human milk probiotic Lactobacillus fermentum CECT5716 reduces the incidence of gastrointestinal and upper respiratory tract infections in infants. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):55-61. doi: 10.1097/MPG.0b013e3182333f18. PMID 21873895
- [Result] Merenstein D, Murphy M, Fokar A, Hernandez RK, Park H, Nsouli H, Sanders ME, Davis BA, Niborski V, Tondu F, Shara NM. Use of a fermented dairy probiotic drink containing Lactobacillus casei (DN-114 001) to decrease the rate of illness in kids: the DRINK study. A patient-oriented, double-blind, cluster-randomized, placebo-controlled, clinical trial. Eur J Clin Nutr. 2010 Jul;64(7):669-77. doi: 10.1038/ejcn.2010.65. Epub 2010 May 19. PMID 20485304